CLINICAL TRIAL: NCT04554745
Title: The Assessment of Cervical Length and Thickness of Cesarean Section Scar as Predictors for Preterm Labor in Patients With Previous Cesarean Section
Brief Title: The Cervical Length and Thickness of Cesarean Section Scar With Preterm Labor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Khairy Ali, Assistant professor, Assiut University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Preterm labor and previous cs
Record Dates: First submitted 2020-09-13; First posted 2020-09-18 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Preterm Labor
MeSH Terms: conditions — Obstetric Labor, Premature | interventions — High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-scared uterus of pregnant women (Other)
  Interventions: Radiation: Ultrasound
- Scared uterus of pregnant women (Other)
  Interventions: Radiation: Ultrasound

INTERVENTIONS:
Radiation: Ultrasound — ultrasound assessment of pregnant women

SUMMARY:
Although the Cesarean section is one of the most common obstetric operations around the world, the World Health Organization recognizes that where cesarean rates are higher than 10%, there is no increase in beneficial maternal and newborn outcomes. some researchers noted that in countries where cesarean rates are above 15%, populations experience higher maternal, infant, and neonatal mortality rates. infants born by cesarean delivery are more likely to require neonatal intensive care unit and have greater respiratory complications, and higher odds for childhood asthma, and obesity.

Preterm is defined as babies born alive before completing 37 weeks of pregnancy.

Preventing Preterm birth is a global priority due to increased risk for neonatal morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

1. singleton pregnant
2. gestational age at 18 weeks
3. previous vaginal or Cesarean section

Exclusion Criteria:

1. twins pregnancy in their second birth
2. previous preterm labor
3. diabetic during the second pregnancy
4. hypertensive during the second pregnancy
5. cigarette use during the second pregnancy
6. congenital anomalies

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 260 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Number of preterm labor in both groups | 6 months

SECONDARY OUTCOMES:
number of babies will enter the neonatal intensive care unit | 6 months
Gestational age at time of delivery | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Abo Al Fadl Elsayed Mohammed, Asst.prof, Study Director — Assiut University
Locations (1):
- Amr, Asyut, Egypt

REFERENCES:
- [Background] Hu HT, Xu JJ, Lin J, Li C, Wu YT, Sheng JZ, Liu XM, Huang HF. Association between first caesarean delivery and adverse outcomes in subsequent pregnancy: a retrospective cohort study. BMC Pregnancy Childbirth. 2018 Jun 28;18(1):273. doi: 10.1186/s12884-018-1895-x. PMID 29954355
- [Background] Urquia ML. Is the association between previous caesarean section and preterm delivery causal? BJOG. 2020 Apr;127(5):618. doi: 10.1111/1471-0528.16099. Epub 2020 Feb 10. No abstract available. PMID 31953981
- [Background] Visser L, Slaager C, Kazemier BM, Rietveld AL, Oudijk MA, de Groot C, Mol BW, de Boer MA. Risk of preterm birth after prior term cesarean. BJOG. 2020 Apr;127(5):610-617. doi: 10.1111/1471-0528.16083. Epub 2020 Feb 24. PMID 31883402
- [Background] Wang M, Kirby A, Gibbs E, Gidaszewski B, Khajehei M, Chua SC. Risk of preterm birth in the subsequent pregnancy following caesarean section at full cervical dilatation compared with mid-cavity instrumental delivery. Aust N Z J Obstet Gynaecol. 2020 Jun;60(3):382-388. doi: 10.1111/ajo.13058. Epub 2019 Sep 12. PMID 31514230
- [Background] Williams CM, Asaolu I, Chavan NR, Williamson LH, Lewis AM, Beaven L, Ashford KB. Previous cesarean delivery associated with subsequent preterm birth in the United States. Eur J Obstet Gynecol Reprod Biol. 2018 Oct;229:88-93. doi: 10.1016/j.ejogrb.2018.08.013. Epub 2018 Aug 11. PMID 30130688
- [Background] Yasseen Iii AS, Bassil K, Sprague A, Urquia M, Maguire JL. Late preterm birth and previous cesarean section: a population-based cohort study. J Matern Fetal Neonatal Med. 2019 Jul;32(14):2400-2407. doi: 10.1080/14767058.2018.1438397. Epub 2018 Feb 21. PMID 29415589
- [Background] Zhang N, Chen H, Xu Z, Wang B, Sun H, Hu Y. Pregnancy, Delivery, and Neonatal Outcomes of In Vitro Fertilization-Embryo Transfer in Patient with Previous Cesarean Scar. Med Sci Monit. 2016 Sep 16;22:3288-95. doi: 10.12659/msm.900581. PMID 27636504
- [Background] Zhang Y, Zhou J, Ma Y, Liu L, Xia Q, Fan D, Ai W. Mode of delivery and preterm birth in subsequent births: A systematic review and meta-analysis. PLoS One. 2019 Mar 14;14(3):e0213784. doi: 10.1371/journal.pone.0213784. eCollection 2019. PMID 30870524